CLINICAL TRIAL: NCT01951209
Title: Prospective Pilot Study of the Effect of Rifaximin on B-Cell Dysregulation in Cirrhosis Due to Chronic Hepatitis C Infection
Brief Title: Pilot Study Of The Effect Of Rifaximin On B-Cell Dysregulation In Cirrhosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment prior to expiration date of unreplaceable blinded investigational product
Sponsor: David E. Kaplan, MD MSc (U.S. Federal Agency)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor-Investigator, David E. Kaplan, MD MSc, GI Staff Physician, Corporal Michael J. Crescenz VA Medical Center
Organization: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 01478
Record Dates: First submitted 2013-09-20; First posted 2013-09-26 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Liver Cirrhosis; Chronic Hepatitis C
Keywords: Human; Hepatitis C; Cirrhosis; B-cell; Rifaximin
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis C, Chronic; Hepatitis C; Fibrosis | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin/Placebo (Experimental): Rifaximin 550mg po bid for 12 weeks followed by crossover to matched placebo po bid x 12 weeks
  Interventions: Drug: Rifaximin; Drug: Placebo
- Placebo/Rifaximin SSD (Experimental): Matched placebo po bid for 12 weeks followed by crossover to Rifaximin 550mg po bid x 12 weeks
  Interventions: Drug: Rifaximin; Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — 550mg orally twice daily for 12 weeks
  Other Names: Rifaximin (Xifaxan)
Drug: Placebo — Matched placebo

SUMMARY:
Hepatitis C is the leading cause of chronic liver disease and cirrhosis in United States veterans. Cirrhosis is associated with impaired antibody responses and increased risk of bacterial infections. We have recently identified that cirrhosis is associated with abnormalities of memory B-cells, cells that make antibodies and help protect against bacterial infections. We have identified that chemicals associated with gut bacteria might play a role in causing these B-cell abnormalities. It is well known that gut bacteria have increased access to the blood in individuals with cirrhosis, a process called bacterial translocation. We hypothesize that reducing bacteria counts in the gut by using poorly-absorbed antibiotics (also known as selective gut decontamination) will partially reverse losses of memory B-cells in cirrhosis by reducing bacterial translocation.

DETAILED DESCRIPTION:
We intend to enroll 18 patients with cirrhosis who do not have hepatic encephalopathy to prospectively evaluate the impact of rifaximin on B-cell phenotype and function. We plan to employ a randomized, double-masked, prospective crossover design to minimize bias. Subjects will be randomized to receive either rifaximin SSD 80mg or a matched placebo once daily for 12 weeks then crossed over to opposite therapy for 12 weeks. Serum and lymphocytes will be collected at baseline and every 4 weeks for in vitro assessment markers of gut microbial translocation and B-cell assays. Stool will be collected at baseline and every 12 weeks for future evaluation of changes of the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Current or prior chronic Hepatitis C infection as documented by detectable HCV RNA in prior 5 years
* Child-Turcotte-Pugh stage A5-B8. Cirrhosis diagnosis may be based on either histological criteria (an previous liver biopsy showing F4/4 or F5-6/6 fibrosis) or clinical criteria (nodular liver on abdominal imaging, splenomegaly, thrombocytopenia, spider telangiectasias, palmar erythema, ascites, varices).
* Platelet count < 175,000/ul
* Subject capable of giving informed consent

Exclusion Criteria:

* Active alcohol use > 20g/d
* Current or planned (within following 6 months) antiviral therapy for hepatitis C
* HIV co-infection
* Diagnosis of overt hepatic encephalopathy
* Current lactulose use
* Exposure to rifaximin, rifampin or rifabutin within 12 months
* History of C. difficile colitis
* History of adverse drug reaction or sensitivity to rifaximin, rifampin or rifabutin or any inactive components of rifaximin
* Pregnancy
* Anemia with hemoglobin < 10g/dl or hematocrit < 30%
* Chronic kidney disease with creatinine > 2.1mg/dl
* Total bilirubin > 3.0g/dl
* Active non-hepatic medical conditions such as congestive heart failure, chronic lung disease requiring oxygen, coronary artery disease with unstable angina
* Requirement for chronic immunosuppressive therapy such as corticosteroids, cyclophosphamide, azathioprine, TNF-alpha antagonists
* Chronic autoimmune diseases such as systemic lupus erythematosus and rheumatoid arthritis
* Post-liver transplantation status or anticipated liver transplantation within 6 months.
* Systemic antimicrobial exposure within 30 days of planned Visit 1

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
Change in CD27+ B-cell frequency | Week 0 (Baseline) to Week 12

SECONDARY OUTCOMES:
Change in basal B-cell activation | Week 0 to Week 12
  5 x 104/well B-cells negatively selected from normal donor PBMC will be cultured in 50% RPMI 1640/50% cirrhotic patient serum for 48 hours. After 48 hours, B-cells will be assessed for activation markers such as HLA-DR geometric mean fluorescence intensity.

OTHER OUTCOMES:
Change in circulating markers of bacterial translocation | Week 0 to Week 12
  Plasma samples will be studied for sCD14 by ELISA, bacterial DNA by rtPCR of 16S ribosomal RNA using established techniques, and Limulus Amebocyte Lysate Assay

CONTACTS AND LOCATIONS:
Overall Officials: David E Kaplan, MD, MSc, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center
Locations (1):
- Philadelphia VA Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified primary data will be made available for verification

REFERENCES:
- [Background] Doi H, Iyer TK, Carpenter E, Li H, Chang KM, Vonderheide RH, Kaplan DE. Dysfunctional B-cell activation in cirrhosis resulting from hepatitis C infection associated with disappearance of CD27-positive B-cell population. Hepatology. 2012 Mar;55(3):709-19. doi: 10.1002/hep.24689. Epub 2012 Jan 19. PMID 21932384